CLINICAL TRIAL: NCT03211689
Title: The Impact of Exercise on Stress, Fatigue, and Quality of Life in Individuals With Primary Immunodeficiency Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockton University (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Kerri Sowers PT, DPT, NCS, Assistant Professor of Health Science, Stockton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010183; IRB00002823 (Other: Nova Southeastern University)
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Primary Immune Deficiency Disorder; Common Variable Immunodeficiency; Specific Antibody Deficiency; Hypergammaglobulinemia
Keywords: Exercise; Stress; Fatigue; Quality of Life
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Hypergammaglobulinemia; Motor Activity; Fatigue | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants will engage in up to 150 minutes of exercise per week, at a level of 11-14 on the Borg Rate of Perceived Exertion scale.
  Interventions: Other: Exercise Program
- Control Group (No Intervention): Participants will continue normal activities, with no new participation in exercise program (may engage in less than 75 minutes of non-structured exercise per week).

INTERVENTIONS:
Other: Exercise Program — Participants will utilize the Physitrack exercise program to engage in up to 150 minutes of exercise at a rating of 11-14 on the Borg Rate of Perceived Exertion scale, per week.
  Arms: Exercise Group

SUMMARY:
This aim of this research project is to determine if low to moderate level exercise can have an impact on stress, fatigue, and quality of life for individuals diagnosed with a primary immunodeficiency disease. This 8-week study will compare participants engaging in a semi-customized, home exercise program (exercise intervention group) to participants performing normal activities (non-exercise control group). This study will track stress, fatigue, and quality of life in individuals with a diagnosis of primary immunodeficiency disease, using standardized questionnaires, journals, and interviews.

DETAILED DESCRIPTION:
This aim of this research project is to determine if low to moderate level exercise can have an impact on stress, fatigue, and quality of life for individuals diagnosed with a primary immunodeficiency disease. Many individuals diagnosed with primary immunodeficiency disease report chronic fatigue and/or pain, which can potentially limit their participation in exercise and physical activities. Research shows that regular exercise can improve both physical and mental health for individuals diagnosed with a chronic medical condition. Exercise is a healthy and low-cost alternative to some medications, and may be an effective addition to the treatment plan for many patients with primary immunodeficiency disease. Research also suggests that low level exercise may be beneficial to immune function, while intense, or prolonged exercise can be harmful. This 8-week study will compare participants engaging in a semi-customized, home exercise program (exercise intervention group) to participants performing normal activities (non-exercise control group). This study will track stress, fatigue, and quality of life, using standardized questionnaires, journals, and interviews. Weekly contact will be made with all participants throughout the 8 weeks of the study. Individuals in the exercise group will be asked to complete up to 150 minutes of exercise, per week, at the 11-14 rating of perceived exertion. Participants who are randomized to the control group will continue their normal activities; they will also be given the opportunity to participate in the exercise program at the end of the 8 week study. To help assess the safety of a low to moderate level exercise program for individuals with primary immunodeficiency disease, this research will track the number of infections, non-planned medical visits, or increased medication usage during the study (compared to 8 weeks prior to the intervention). This research will help provide valuable information about the safety and effectiveness of an exercise program for individuals with a primary immunodeficiency disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Physician diagnosis of a primary immunodeficiency disease (as evidenced by physician letter or medical documentation/report)
* Willingness to participate in eight-week exercise program

Exclusion Criteria:

* Current participation in a structured exercise program for greater than 75 minutes per week
* Any medical condition that prevents participation in a low to moderate level exercise program (such as, but not limited to, uncontrolled asthma, unstable cardiac condition, acute orthopedic injury which requires restricted activities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Short Form 36 version 2 | Change during 8 weeks
  Measure of quality of life.

SECONDARY OUTCOMES:
Infection Incidence | Change from 8 weeks prior to the start of study to the 8 weeks during the study
  Measure of number of infections that have occurred
Unplanned use of medical provider | Change from 8 weeks prior to the start of the study to the 8 weeks during the study.
  Number of unplanned visits to a medical provider
Fatigue Impact Scale | Change during 8 weeks
  Measure of fatigue.
Exercise Benefits/Barriers Scale | Change during 8 weeks
  Measure of perceptions about exercise.
Perceived Stress Scale 10 | Change during 8 weeks
  Measure of stress.
Self-efficacy for Exercise Scale | Change during 8 weeks
  Measure about ability to comply with exercise program
Subjective Exercise Experience Scale | Change during 8 weeks
  Measures perceptions about participation in an exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Sowers, PT, DPT, NCS, Principal Investigator — Stockton University
Locations (1):
- Stockton University, Galloway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No